CLINICAL TRIAL: NCT04870840
Title: Proton Image-Guided Radiation Assignment for Therapeutic Escalation Via Selection of Locally Advanced Head and Neck Cancer Patients [PIRATES]
Brief Title: Image-guided Proton Therapy for the Treatment of Locally Advanced Unresectable Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0467; NCI-2020-04072 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0467 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-23; First posted 2021-05-04 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma; Locally Advanced Hypopharyngeal Squamous Cell Carcinoma; Locally Advanced Laryngeal Squamous Cell Carcinoma; Locally Advanced Nasopharyngeal Squamous Cell Carcinoma; Locally Advanced Oral Cavity Squamous Cell Carcinoma; Locally Advanced Oropharyngeal Squamous Cell Carcinoma; Malignant Posterior Tongue Neoplasm; Stage II Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage II Hypopharyngeal Carcinoma AJCC v8; Stage II Laryngeal Cancer AJCC v8; Stage II Nasopharyngeal Carcinoma AJCC v8; Stage II Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Nasopharyngeal Carcinoma AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Unresectable Head and Neck Squamous Cell Carcinoma; Unresectable Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Carcinoma; Carcinoma | interventions — Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (proton therapy) (Experimental): Patients undergo radiation therapy QD 5 days a week (Monday through Friday) for the first 18 days and then BID for 15 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Proton Beam Radiation Therapy — Undergo radiation therapy
  Other Names: PBRT; Proton Radiation Therapy; Radiation, Proton Beam
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects of image-guided hyper-fractioned proton therapy in treating patients with head and neck cancer that has spread to nearby tissue or lymph nodes (locally advanced) and cannot be removed by surgery (unresectable). Radiation therapy uses high energy protons to kill tumor cells and shrink tumors. The change in dose radiation frequency and dose investigated in this study may help to better control the tumor and prevent it from coming back or growing. The goal of this study is to test a new radiation schedule that administers more radiation to the tumor tissue using image guided proton therapy for patients that have a high risk of having a tumor recurrence (the tumor comes back after treatment).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety & feasibility of image guided mid-treatment hyper-fractioned dose-escalation with proton therapy and identify the maximum tolerable dose (MTD) for the treatment of locally advanced human papillomavirus (HPV) negative head and neck cancer.

OUTLINE:

Patients undergo radiation therapy once daily (QD) 5 days a week (Monday through Friday) for the first 18 days and then twice daily (BID) for 15 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 8 weeks, 3, 6, 9, and 12 months in the first year after radiation therapy, every 4 months in the second year after radiation therapy, and then every 9 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven diagnosis of squamous cell carcinoma of head and neck cancer originating in the oropharynx, hypopharynx, larynx, oral cavity (base of tongue) or nasopharynx. Clinical evidence should be documented, and may consist of imaging, endoscopic evaluation, palpation, and should be sufficient to estimate the image tumor characteristic of the primary tumor
* Negative for HPV by p16 immunohistochemistry (IHC) or in situ hybridization (ISH)
* Inoperable locally advances disease, i.e. stage >= III and T stage >= 2
* The primary radiotherapy, either in combination with chemotherapy or not, with curative intent
* No head and neck surgery of the primary tumor or lymph nodes except for incisional or excisional biopsies
* Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2
* For females of child-bearing age, a negative pregnancy test

Exclusion Criteria:

* Patients who have undergone definitive resection of their primary or nodal disease as well as any chemotherapy or radiation therapy for their head and neck squamous cell carcinoma (HNSCC)
* Patient that refuse or are unable to stop smoking and/or consuming alcohol during and after radiotherapy. In addition, patients that refuse or fail tobacco and alcohol blood test
* Patients that have no detectable no tumor in both the primary site and lymph nodes at week 4 in treatment, because there will not be a volume to boost
* Patients unable or unwilling to give written, informed consent or to undergo magnetic resonance imaging (MRI) imaging
* Women of childbearing potential (a woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]). Male partners must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study
* Patients unable to tolerate intravenous contrast for both computed tomography (CT) and MRI, having an estimated glomerular filtration rate (GFR) < 60 ml/min/1.73 m^2 or any contraindications to gadolinium-based contrast agents
* Contraindications to iron supplementation include hemochromatosis, colitis, history of gastrointestinal (GI) bleeds, alcoholism, or liver disease. Ferumoxytol is contraindicated in patients with evidence of iron overload and/or known hypersensitivity to Feraheme or any of its components. Consequently, we will plan to exclude patients who have symptoms or signs that might be caused by iron overload. These include patients with (unexplained): arthritis (including premature osteoarthritis), congestive heart failure or cardiomyopathy, adult-onset diabetes, secondary hypogonadism, increased skin pigmentation, or patients with persistently elevated serum ferritin not explained by an underlying inflammatory/systemic disease, unless these patients demonstrate a fasting transferrin saturation =< 0.45
* Patients with any evidence of iron overload on pre-imaging laboratory studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of severe unacceptable local adverse events which are radio therapeutically attributable | Up to 6 months after radiation therapy
  Specifically, Common Terminology Criteria for Adverse Events (CTCAE) version 5 grade 4 mucositis, dermatitis or aspiration that does not resolve to a grade =< 3 in 3 months, and CTCAE version 5 grade >= 3 myelopathy, and/or osteonecrosis. Summary statistics, including mean, standard deviation and 95% confidence interval will be used to describe safety data. Toxicity will be tabulated and summarized by grade and type.

SECONDARY OUTCOMES:
Incidence of grade 3 toxicity | At 3-6 months after radiation therapy
  Specifically, CTCAE version 5 grade 3 mucositis, dermatitis, aspiration, dysphagia, hearing impaired, xerostomia, weight loss, trismus, hoarseness, oropharyngeal pain. Summary statistics, including mean, standard deviation and 95% confidence interval will be used to describe safety data. Toxicity will be tabulated and summarized by grade and type. Radiation induced side effect (RISE) rate will be summarized by frequency, standard deviation and 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton D Fuller, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] van Dijk LV, Frank SJ, Yuan Y, Gunn B, Moreno AC, Mohamed ASR, Preston KE, Qing Y, Spiotto MT, Morrison WH, Lee A, Phan J, Garden AS, Rosenthal DI, Langendijk JA, Fuller CD. Proton Image-guided Radiation Assignment for Therapeutic Escalation via Selection of locally advanced head and neck cancer patients [PIRATES]: A Phase I safety and feasibility trial of MRI-guided adaptive particle radiotherapy. Clin Transl Radiat Oncol. 2021 Nov 11;32:35-40. doi: 10.1016/j.ctro.2021.11.003. eCollection 2022 Jan. PMID 34841093
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT04870840/ICF_000.pdf